CLINICAL TRIAL: NCT05012436
Title: A Study to Evaluate the Pharmacokinetics and Safety Following a Single Oral Dose of YHD1119 in Subjects With Renal Impairment and Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of YHD1119 in Subjects With Renal Impairment and Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YHD1119-107
Record Dates: First submitted 2021-07-27; First posted 2021-08-19 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteer; Renal Impairments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YHD1119 75mg, 150mg NF (Experimental): CLcr (mL/min/1.73m2) >= 60 Period 1 : YHD1119 75 mg Period 2 : YHD1119 150 mg NF
  Interventions: Drug: YHD1119 75mg
- YHD1119 75mg (Experimental): 60 > CLcr (mL/min/1.73m2) >= 30 Period 1 : YHD1119 75 mg Period 2 : NA
  Interventions: Drug: YHD1119 75mg

INTERVENTIONS:
Drug: YHD1119 75mg — A single oral dose
  Other Names: YHD1119 150mg NF

SUMMARY:
The purpose of this trial is to compare the pharmacokinetic characteristics and safety of YHD1119(Pregabalin SR 75mg) and YHD1119(Pregabalin SR 150mg) in subjects with renal impairment and healthy subjects. YHD1119 is sustained-release (SR) formulation which is made by Yuhan Corporation. Primary endpoints are Cmax and AUClast and secondary endpoints are AUCinf,Tmax, t1/2, CL/F and V/F.

ELIGIBILITY:
Inclusion Criteria:

* 19~75 years old, healthy volunteers and renal impairments
* eGFR >= 60mL/min/1.73m2
* 60 mL/min/1.73m2 > eGFR >= 30mL/min/1.73m2
* written informed consent

Exclusion Criteria:

* AST or ALT > 1.5 * Upper normal range
* Total bilirubin > 1.5 * Upper normal range
* Blood CPK > 1.5 * Upper normal range
* Total Cholesterol >1.5 * Upper normal range
* Woman who is pregnant or lactating
* Patients who are difficult to participate in cinical trials judged by Investigators
* have participated in other clinical trials within 180 days before IP intake

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-24 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour
AUClast | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour

SECONDARY OUTCOMES:
AUCinf | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour
Tmax | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour
t1/2 | 0,1,2,3,4,5,6,8,10,12,14,24,48,72hour
CL/F | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour
V/F | 0,1,2,3,4,5,6,8,10,12,14,24,48,72 hour

CONTACTS AND LOCATIONS:
Overall Officials: SeungHoon Han, Principal Investigator — The Catholic University of Korea; Hyounggyoon Yoo, Principal Investigator — CHA University
Locations (2):
- South Korea (2):
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park M, Choi S, Han S, Shin W, Kim A, Han S, Kim B, Lim Y, Yoo H. Pharmacokinetic properties of a new sustained-release pregabalin tablet in subjects with reduced renal function. Transl Clin Pharmacol. 2023 Dec;31(4):226-237. doi: 10.12793/tcp.2023.31.e20. Epub 2023 Dec 20. PMID 38197000